CLINICAL TRIAL: NCT03571685
Title: A Prospective, Open Label, Quasi-Experimental Study of Adult Patients With Schizophrenia or Schizoaffective Disorder Within Five Years of Diagnosis Who Will Receive SEEC Intervention
Brief Title: Sustainable Early Episode Clinic Study (SEEC)
Acronym: SEEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-08A
Record Dates: First submitted 2018-03-01; First posted 2018-06-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: This is an open label, quasi-experimental study of adult patients with Schizophrenia or Schizoaffective Disorder within five years of diagnosis who are receiving SEEC intervention in phases. Approximately 50 patients will be enrolled in the study. Caregivers who would like to participate will also be included. Patients will be followed prospectively over the study period up to 36 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sustainable Early Episode Clinic Model of Care (Experimental): The model of care given in the sustainable early episode clinic study, provides early intense intervention, with an ongoing maintenance phase in an outpatient setting.
  Interventions: Behavioral: Sustainable Early Episode Clinic Model of Care

INTERVENTIONS:
Behavioral: Sustainable Early Episode Clinic Model of Care — The first 8 weeks is the education phase. Participants attend classes every week for up to 6 hours. From 9 weeks to 10 months participants attend classes for 5 hours every other week. Based on individual progress. Participants can move to the maintenance phase. This phase provides minimal intervention but ongoing support/evaluation.

SUMMARY:
The purpose of this study is to describe relapse rates among participants receiving services in the SEEC program high intensity resource use. For purposes of this study, relapse will be defined as: Psychiatric hospitalization; Psychiatric emergency department visits; Ambulatory acute services (Partial Hospitalization Program, Intensive Outpatient Program, Crisis House stay).

DETAILED DESCRIPTION:
Schizophrenia is a severe mental illness that is one of the leading causes of long-term disability in the world. Recognizing the need for improved early treatment for participants diagnosed with Schizophrenia or Schizoaffective Disorder, a model was created for a "sustainable early episode clinic, SEEC." The goal of the SEEC model is to provide early intense intervention in 3 phases, with an ongoing maintenance phase, enabled by technology, resulting in improved participant outcomes and reduced long-term economic and social burden of schizophrenia. This study will last for up to a 36-month period.

ELIGIBILITY:
Inclusion Criteria - Participants

* Participants must be at least 18 years or older
* Participants within 5 years of a clinical diagnosis of Schizophrenia or Schizoaffective disorder made by a clinician with understanding of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for these disorders
* Participants must be able to speak, read, and understand English
* Participants must sign an informed consent form

Inclusion Criteria - Caregivers

* Caregivers must be 18 years or older Caregivers must also be willing to attend the multi-family psychoeducation group series (Phase I)
* Caregivers must be willing to participate in monthly family therapy and/or monthly phone contact with staff for the duration of the study
* Caregivers must sign informed consent form

Exclusion Criteria - Participants

* Co-occurring developmental disabilities
* Receiving electroconvulsive therapy
* Primary substance use disorder
* On permanent conservatorship
* Unable to complete baseline assessments due to acuity of psychiatric symptoms

Exclusion Criteria - Caregivers

* Caregivers who refuse to participate in the psychoeducation series of Phase 1
* Caregivers who refuse monthly family therapy/phone contact with staff will be excluded
* Caregiver is mentally or physically incapable of adequately performing the required study procedures, as determined by treatment team
* Caregiver is an employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employee or the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
High Intensity Service Utilization Rate | Baseline up to 36 months
  The rate of high intensity service utilization that is count per unit of time for mental health services will be reported. It is evaluated as the number of psychiatric hospitalizations, behavioral health emergency department visits, and number of times referred to a partial hospitalization program (PHP), intensive outpatient program (IOP), or Crisis Unit.

SECONDARY OUTCOMES:
Overall Healthcare Utilization Rate | Baseline up to 36 months
  Overall healthcare utilization rate that is count per unit of time of the healthcare resources which were utilized by the participants over over the time will be reported.
Change from Baseline in Clinician-Rated Dimensions of Psychosis Symptom and Severity (CRDPSS) Scale | Baseline up to 36 months
  The CRDPSS is an 8 item measure that assesses the severity of mental health symptoms that are important across psychotic disorders including:
  Delusions, hallucinations, disorganized speech, abnormal psycho-motor behavior, negative symptoms, impaired cognition, depression and mania. Each item on the measure is rated on a 5 point scale with a symptom specific definition of each rating level: 0 = none, 1= equivocal, 2= present but mild, 3= present and moderate, 4= present and severe. Total Score is taken as summation. High score indicates worsening of symptoms.
Change from Baseline in Clinical Global Impressions Scale (CGI-S) | Baseline up to 36 months
  The CGI-S measures illness severity and is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (among the most severely ill participants).
Change from Baseline in Personal and Social Performance (PSP) Scale | Baseline up to 36 months
  The PSP has 4 domains of functioning considered in this scale: (a) Socially useful activities including work and study, (b) Personal & Social Relationships, (c) Self Care (d) Disturbing and aggressive behaviors. All rated from absent, mild, manifest, marked, severe and very severe. Scores of 1-30 reflect functioning so poor that the participant requires intensive support of supervision. 31-70 varying degree of difficulties 71-100 reflect only mild difficulties.
Change from Baseline in Perceived Family Burden Scale (PFBS) | Baseline up to 36 months
  The purpose of the PFBS scale is to measure the burden of schizophrenia on the family of a participant. It is a 24-item questionnaire rated on a 5 point Likert type scale: 0 = the behavior isn't present and doesn't bother the relative, 1 = the behavior is present and doesn't bother the relative, 2 = the behavior is present and bothers the relative "a little", 3 = the behavior is present and bothers the relative "considerably", 4 = the behavior is present and bothers the relative "a great deal". High score indicates worsening of burden.
Heinrichs-Carpenter Quality of Life Scale (QLS) | Baseline up to 36 months
  The QLS is used to evaluate defect symptoms and impaired functioning in non-hospitalized schizophrenic participants. It is a 21-item scale providing information on symptoms and functioning in the preceding 4 weeks. Each item is rated on 7 point scale. A sub scale score is being used in 4 sections ranging from 0-56. Low score represents worse functioning. Then a total score is taken by adding the 4 sections. Range of possible scores, 0-126. Lower sub scale scores and total scores indicates lower quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (1):
- Sharp Outpatient Behavioral Health Clinic, San Diego, California, United States